CLINICAL TRIAL: NCT01327989
Title: STAR: Solitaire FR Thrombectomy for Acute Revascularisation
Brief Title: Solitaire FR Thrombectomy for Acute Revascularisation
Acronym: STAR
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Collaborators: ev3 International (Industry)
Responsible Party: Sponsor
Other Study IDs: ev3-02-2010
Record Dates: First submitted 2010-10-12; First posted 2011-04-04 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-10

CONDITIONS: Stroke, Acute
Keywords: Solitaire FR Device; Mechanical Thrombectomy; Recanalization; Brain artery recanalization; Neurovascular intervention; Interventional Neuroradiology; STAR; Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Solitaire™ FR device: Eligible subjects treated with the Solitaire™ FR device.
  Interventions: Device: Solitaire™ FR device

INTERVENTIONS:
Device: Solitaire™ FR device — Mechanical Thrombectomy

SUMMARY:
The objective of this study was to obtain prospective clinical data on the safety and efficacy of the Solitaire™ FR device for patients diagnosed with acute ischemic stroke.

DETAILED DESCRIPTION:
The Study was a multi-center, single-arm, prospective, observational evaluation. The Solitaire™ FR Device has been certified for CE mark. This protocol evaluated the safety and efficacy of the Solitaire™ FR Device when used in routine practice and according to its Instructions for Use.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's legally authorized representative has signed and dated an Informed Consent Form
2. Age ≥ 18 and < 85
3. Clinical signs consistent with acute ischemic stroke
4. Thrombolysis in Cerebral Infarction (TICI) 0 or TICI 1 flow in the proximal anterior intracranial vasculature (M1 or M2 of Middle Cerebral Artery (MCA), Internal Carotid Artery (ICA) intracranial, Internal Carotid Artery (ICA) terminal)
5. Presentation within 8 hours of stroke onset according to local stroke protocol
6. If stroke presentation within 4.5 hours, one of these conditions can be met:

   * Bridging protocol (starting intravenous and continuing with intra-arterial) (Up to maximum 0.9 mg/kg)
   * Failed intravenous thrombolysis
   * Direct Intra-arterial treatment (according to institution guidelines)
7. Subject is willing to conduct follow-up visits.
8. National Institutes of Health Stroke Scale (NIHSS) ≥ 8 and ≤ 30
9. Modified Rankin Scale (mRS) ≤ 2 prior to stroke onset

Exclusion Criteria:

1. Females who are pregnant or lactating
2. Known serious sensitivity to radiographic contrast agents
3. Neurological signs that are rapidly improving prior to or at time of treatment
4. Current participation in another investigational drug or device study
5. Life expectancy of less than 90 days
6. National Institutes of Health Stroke Scale (NIHSS) > 30 or coma
7. Uncontrolled hypertension defined as systolic blood pressure > 185 or diastolic blood pressure > 110 that cannot be controlled except with continuous parenteral antihypertensive medication
8. Use of warfarin anticoagulation with International Normalised Ratio (INR) > 3.0
9. Platelet count < 30,000
10. Glucose < 400 mg/dL
11. Previous stroke within 30 days
12. Time of symptom onset unknown
13. Seizure at the onset of stroke
14. Myocardial infarction or infection (sepsis or endocarditis)
15. Arterial tortuosity that would prevent the device from reaching the target vessel
16. Known hypersensitivity to nickel-titanium

    Imaging Exclusion Criteria:
17. Angiographic evidence of carotid dissection, complete cervical carotid occlusions, or vasculitis
18. Stenosis proximal to thrombus site that may preclude safe recovery of the device
19. Brain computed tomography (CT) with signs of hemorrhage, arteriovenous venous malformations, or aneurysm
20. Early ischemic changes greater than 1/3 of the middle cerebral artery (MCA) territory or according to brain computed tomography (CT) Alberta Stroke Program Early CT (ASPECT) score ≤ 6 or according to magnetic resonance diffusion weighted imaging (MR DWI) ASPECT score <5

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having clinical signs and imaging criteria consistent with acute ischemic stroke who presented within 8 hours of stroke symptoms onset with the study device were considered for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Mendes Pereira, Dr, Principal Investigator — HUG Geneva; Jan Gralla, Dr, Principal Investigator — Inselspital University Hospital of Bern
Locations (2):
- Switzerland (2):
  - Inselspital University Hospital of Bern, Bern
  - Hôpitaux Universitaires de Genève (HUG), Geneva

REFERENCES:
- [Derived] Raychev R, Saver JL, Jahan R, Nogueira RG, Goyal M, Pereira VM, Gralla J, Levy EI, Yavagal DR, Cognard C, Liebeskind DS. The impact of general anesthesia, baseline ASPECTS, time to treatment, and IV tPA on intracranial hemorrhage after neurothrombectomy: pooled analysis of the SWIFT PRIME, SWIFT, and STAR trials. J Neurointerv Surg. 2020 Jan;12(1):2-6. doi: 10.1136/neurintsurg-2019-014898. Epub 2019 Jun 25. PMID 31239326
- [Derived] Coutinho JM, Liebeskind DS, Slater LA, Nogueira RG, Clark W, Davalos A, Bonafe A, Jahan R, Fischer U, Gralla J, Saver JL, Pereira VM. Combined Intravenous Thrombolysis and Thrombectomy vs Thrombectomy Alone for Acute Ischemic Stroke: A Pooled Analysis of the SWIFT and STAR Studies. JAMA Neurol. 2017 Mar 1;74(3):268-274. doi: 10.1001/jamaneurol.2016.5374. PMID 28097310
- [Derived] Menon BK, Almekhlafi MA, Pereira VM, Gralla J, Bonafe A, Davalos A, Chapot R, Goyal M; STAR Study Investigators. Optimal workflow and process-based performance measures for endovascular therapy in acute ischemic stroke: analysis of the Solitaire FR thrombectomy for acute revascularization study. Stroke. 2014 Jul;45(7):2024-9. doi: 10.1161/STROKEAHA.114.005050. Epub 2014 May 15. PMID 24876244
- [Derived] Almekhlafi MA, Davalos A, Bonafe A, Chapot R, Gralla J, Pereira VM, Goyal M; STAR Registry Investigators. Impact of age and baseline NIHSS scores on clinical outcomes in the mechanical thrombectomy using solitaire FR in acute ischemic stroke study. AJNR Am J Neuroradiol. 2014 Jul;35(7):1337-40. doi: 10.3174/ajnr.A3855. Epub 2014 Feb 20. PMID 24557701
- [Derived] Pereira VM, Gralla J, Davalos A, Bonafe A, Castano C, Chapot R, Liebeskind DS, Nogueira RG, Arnold M, Sztajzel R, Liebig T, Goyal M, Besselmann M, Moreno A, Moreno A, Schroth G; the STAR Investigators. Prospective, multicenter, single-arm study of mechanical thrombectomy using Solitaire Flow Restoration in acute ischemic stroke. Stroke. 2013 Oct;44(10):2802-7. doi: 10.1161/STROKEAHA.113.001232. Epub 2013 Aug 1. PMID 23908066

RESULTS

PARTICIPANT FLOW:
Groups:
- Solitaire™ FR Device: Eligible subjects treated with the Solitaire™ FR device.
  Solitaire™ FR device
Period: Overall Study
Arm/Group | Solitaire™ FR Device
Started | 202
Completed | 188
Not Completed | 14

BASELINE CHARACTERISTICS:
Population: Pre-stroke mRS scores are missing for 24 subjects as it was not recorded or determinable.
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (12.5)
Gender [Count of Participants; unit: Participants]
  Female | 122
  Male | 80
Modified Rankin Scale (mRS) [Median (Inter-Quartile Range); unit: Scores on a scale] — The mRS measures degree of disability. (0 No symptoms at all, 1 No significant disability despite symptoms; able to carry out all usual duties and activities, 2 Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance, 3 Moderate disability; requiring some help, but able to walk without assistance, 4 Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance, 5 Severe disability; bedridden, incontinent and requiring constant nursing care and attention, 6 Dead)
  Scores on a scale | 0.0 [0.0 to 3.0]

OUTCOME MEASURES:

1. Primary Outcome: Arterial Recanalization of the Occluded Target Vessel Measured by Thrombolysis in Cerebral Infarction (TICI) Score Equal or Superior to 2b Following the Use of the Study Device.
Description: Thrombolysis in Cerebral Infarction (TICI) score
  Grade 0- No perfusion Grade 1- Penetration with Minimal Perfusion Grade 2- Partial Perfusion Grade 2a- Only partial filling (<2/3) of the entire vascular territory is visualized Grade 2b - Complete filling of all of the expected vascular territory is visualized, but the filling is slower than normal Grade 3- Complete Perfusion
Time Frame: Immediately post procedure
Population: Due to insufficient imaging, the Core Lab was able to evaluate data from 190 subjects.
Measure: Number; unit: percentage of particpants
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 190
percentage of particpants | 84.2

2. Secondary Outcome: Time to Achieve Revascularization - Groin Stick to Initial Angiogram and Final Solitaire™ FR Angiogram
Description: Time from groin stick to initial angiogram and final Solitaire™ FR angiogram with Thrombolysis in Cerebral Infarction (TICI) score 2b or 3 flow
  Thrombolysis in Cerebral Infarction (TICI) score
  Grade 0- No perfusion Grade 1- Penetration with Minimal Perfusion Grade 2- Partial Perfusion Grade 2a- Only partial filling (<2/3) of the entire vascular territory is visualized Grade 2b - Complete filling of all of the expected vascular territory is visualized, but the filling is slower than normal Grade 3- Complete Perfusion
Time Frame: During procedure
Population: Unavailability of data contributed to fewer subjects analyzed compared to the cohort sample size.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 194
Minutes | 29 (27)

3. Secondary Outcome: Time to Achieve Revascularization - After First Ipsilateral Angiogram to Final Solitaire™ FR Angiogram
Description: Time after first ipsilateral angiogram to final Solitaire™ FR angiogram with Thrombolysis in Cerebral Infarction (TICI) score 2b or 3 flow
  Thrombolysis in Cerebral Infarction (TICI) score
  Grade 0- No perfusion Grade 1- Penetration with Minimal Perfusion Grade 2- Partial Perfusion Grade 2a- Only partial filling (<2/3) of the entire vascular territory is visualized Grade 2b - Complete filling of all of the expected vascular territory is visualized, but the filling is slower than normal Grade 3- Complete Perfusion
Time Frame: During Procedure
Population: Unavailability of data contributed to fewer subjects analyzed compared to the cohort sample size.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 201
Minutes | 37.2 (57.7)

4. Secondary Outcome: Good Neurological Condition
Description: Good neurological outcome (GNO), as defined in the protocol, is a modified Rankin Scale (mRS) score of less than or equal to 2, or National Institutes of Health Stroke Scale (NIHSS) score 0-1, or NIHSS score improvement of 10 points or more from the pre-procedure evaluation
Time Frame: 90 Days
Population: Unavailability of data contributed to fewer subjects analyzed compared to the cohort sample size.
Measure: Number; unit: percentage of particpants
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 169
percentage of particpants | 88.2

5. Secondary Outcome: Rate of Morbidity
Time Frame: 90 Days
Measure: Number; unit: percentage of particpants
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 202
percentage of particpants | 8.4

6. Secondary Outcome: Rate of Mortality
Time Frame: 90 Days
Measure: Number; unit: percentage of particpants
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 202
percentage of particpants | 6.9

7. Secondary Outcome: Incidence of Symptomatic Intracranial Hemorrhage
Description: Symptomatic intracranial hemorrhage, defined as any parenchymal hematoma 1 (PH1), parenchymal hematoma 2 (PH2), intraparenchymal hemorrhage remote from the ischemic field (RIH), intraventricular hemorrhage (IVH), and subarachnoid hemorrhage (SAH) associated with a decline in National Institutes of Health Stroke Scale (NIHSS) ≥ 4 within 24 hrs.
  PH1 - Hematoma within ischemic field with some mild space occupying effect but involving ≤ 30% PH2 - Hematoma within ischemic field with space-occupying effect involving > 30% of the infarcted area RIH - Any intraparenchymal hemorrhage remote from the ischemic field IVH - Intraventricular hemorrhage SAH - Subarachnoid hemorrhage
Time Frame: 24 hours
Measure: Number; unit: percentage of particpants
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 202
percentage of particpants | 1.5

8. Secondary Outcome: Immediate Flow Reperfusion
Description: Immediate reperfusion observed when the Solitaire™ FR device is deployed within the thrombus - Thrombolysis in Cerebral Infarction (TICI) score 2b or 3.
  Grade 0- No perfusion Grade 1- Penetration with Minimal Perfusion Grade 2- Partial Perfusion Grade 2a- Only partial filling (<2/3) of the entire vascular territory is visualized Grade 2b - Complete filling of all of the expected vascular territory is visualized, but the filling is slower than normal Grade 3- Complete Perfusion
Time Frame: procedure
Population: Due to insufficient imaging, the Core Lab was able to evaluated data from 190 subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 190
percentage of participants | 11.6

9. Primary Outcome: Incidence of Device-related and Procedure-related Serious Adverse Events (SAEs).
Description: Device-related and procedure-related Serious Adverse Events (SAEs). A clinically significant procedure complication is defined as a decline in NIHSS of ≥4 or access vessel complication requiring surgery or blood transfusion.
Time Frame: 90 Days
Measure: Number; unit: percentage of events
Arm/Group | Solitaire™ FR Device
Number analyzed (Participants) | 202
percentage of events | 7.4

ADVERSE EVENTS:
Time Frame: 90 Days
Description: Independent Clinical Events Committee (CEC) provided independent, unbiased and consistent adjudication for all reportable adverse events.
Arm/Group | Solitaire™ FR Device
Serious Adverse Events (participants affected / at risk) | 59/202
Other Adverse Events (participants affected / at risk) | 143/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solitaire™ FR Device (N=202)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Gallstone ileus (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Catheter site haematoma (General disorders) | 2 (2)
Death (General disorders) | 2 (2)
Thrombosis in device (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 1 (1)
Heart rate irregular (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Pseudomonas test positive (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain oedema (Nervous system disorders) | 3 (3)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 6 (6)
Coma (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
Intracranial artery dissection (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4)
Neurological decompensation (Nervous system disorders) | 3 (3)
Subarachnoid haemorrhage (Nervous system disorders) | 4 (4)
Syncope (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Delirium tremens (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1)
Cranioplasty (Surgical and medical procedures) | 1 (1)
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1)
Heart valve replacement (Surgical and medical procedures) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Vascular dissection (Vascular disorders) | 2 (2)
Vessel perforation (Vascular disorders) | 1 (1)
Aspiration bronchial (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solitaire™ FR Device (N=202)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 10 (10)
Cardiac failure (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1)
Tongue haematoma (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Device leakage (General disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Application site eczema (General disorders) | 1 (1)
Device difficult to use (General disorders) | 2 (3)
Unevaluable event (General disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1)
Bacterial prostatitis (Infections and infestations) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 7 (7)
Secondary syphilis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 14 (14)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Aspiration bronchial (Investigations) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Thyroid function test abnormal (Investigations) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
CREST syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Basilar artery stenosis (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 2 (2)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 34 (36)
Cerebral thrombosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cerebrovascular spasm (Nervous system disorders) | 3 (3)
Convulsion (Nervous system disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 3 (3)
Haemorrhagic transformation stroke (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 3 (3)
Intracranial artery dissection (Nervous system disorders) | 4 (4)
Ischaemic stroke (Nervous system disorders) | 2 (2)
IVth nerve paresis (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5)
Syncope (Nervous system disorders) | 1 (1)
Tonic convulsion (Nervous system disorders) | 1 (1)
Vascular headache (Nervous system disorders) | 1 (1)
Vertebral artery occlusion (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Apathy (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Post stroke depression (Psychiatric disorders) | 2 (2)
Leukocyturia (Renal and urinary disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory fremitus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Air embolism (Vascular disorders) | 3 (3)
Aortic arteriosclerosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 13 (13)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vascular dissection (Vascular disorders) | 3 (3)
Vasospasm (Vascular disorders) | 54 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician shall not make any publication without providing Sponsor 60 days notice.If Sponsor determines that the proposed publication contains confidential information, Sponsor may require the delay of publication for a period of time not to exceed 90 days and may require that any confidential information be removed from the publication. Sponsor may also require Physician to delay publication until any factual errors or inaccuracies in the publication are corrected.